CLINICAL TRIAL: NCT04423809
Title: Impact of Burden in Caregivers of Patients Hospitalized for a Psychotic Episode: a Multicenter Study
Acronym: AFP
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Januel, head of the clinical research unit, Centre hospitalier de Ville-Evrard, France
Other Study IDs: 2014-A01499-38
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: The Objective of Our Study is to Assess and Take Into Account Early on the Suffering of Family Members
Keywords: Psychiatry Nurse Burden Caregiver
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- caregivers of adult patients hospitalized in psychiatry: a face-to-face interview with a nurse and self-assessment scales.
  Interventions: Other: clinical assessment

INTERVENTIONS:
Other: clinical assessment — assessment of caregivers suffering when a family member is hospitalized
  Other Names: Interview

SUMMARY:
Family support is a positive predictor for psychiatric patients. For example, since the 1980s, it has been shown that family psychoeducation improves patient adherence to care and statistically decreases patient relapse and hospitalization rates by half, resulting in lower care costs. Yet, the stress of hospitalizing a patient, seeing the feelings of shame or guilt of caregiver and the impact on their quality of life are rarely taken into account by caregivers during the first weeks hospitalization in a patient's psychiatry.

Barrelet emphasizes the importance of organizing the meeting in the first hours of hospitalization with the family in order to strengthen the alliance, to improve communication.

ELIGIBILITY:
Inclusion Criteria:

* Family members or relatives
* Over 18 years
* Having a relative

  * First hospitalized in psychiatry or hospitalized in psychiatry within 5 years
  * Over 18 years of age
  * Psychotic episode
  * Having been informed of their participation in this study
* In regular contact with the patient prior to hospitalization, at least 4 hours per week.
* French language
* Signed written informed consent.

Exclusion Criteria:

-Psychiatric pathology of another family member than the hospitalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: caregiver of patient hospitalised in psychiatry
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies-Depression scale | at patient admission
  is a simple tool for assessing depressive symptomatology for the general population

SECONDARY OUTCOMES:
Zarit burden inventory | at patient admission
  to assess burden
Short form 36 | at patient admission
  To assess quality of life
Semi-directional interview | At patient admission
  It consists of five items: subjective feeling, quality of life, social life, mood of the caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de recherche clinique, Neuilly-sur-Marne, Île-de-France Region, France